CLINICAL TRIAL: NCT02851485
Title: Open-label Study to Compare the Bioavailability of an Oral Tablet of GLPG1972 Relative to an Oral Solution After Single-dose Intake in Healthy Subjects and to Evaluate the Effect of Food on the Oral Tablet
Brief Title: Bioavailability Study With GLPG1972
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Galapagos NV (Industry)
Collaborators: PRA Health Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: GLPG1972-CL-103
Record Dates: First submitted 2016-07-28; First posted 2016-08-01 (Estimated); Last update posted 2016-10-04 (Estimated); Status verified 2016-05

CONDITIONS: Osteoarthritis
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- GLPG1972 600 mg oral solution fasted (Experimental): 600 mg GLPG1972 administered as oral solution after overnight fasting
  Interventions: Drug: GLPG1972 600 mg oral solution fasted
- GLPG1972 600 mg oral tablet fasted (Experimental): 600 mg GLPG1972 administered as oral tablet after overnight fasting
  Interventions: Drug: GLPG1972 600 mg oral tablet fasted
- GLPG1972 600 mg oral tablet fed (Experimental): 600 mg GLPG1972 administered as oral tablet after a high-fat high-calorie breakfast
  Interventions: Drug: GLPG1972 600 mg oral tablet fed

INTERVENTIONS:
Drug: GLPG1972 600 mg oral solution fasted — dosing after overnight fasting
  Arms: GLPG1972 600 mg oral solution fasted
Drug: GLPG1972 600 mg oral tablet fasted — dosing after overnight fasting
  Arms: GLPG1972 600 mg oral tablet fasted
Drug: GLPG1972 600 mg oral tablet fed — dosing after high-fat high-calorie breakfast
  Arms: GLPG1972 600 mg oral tablet fed

SUMMARY:
This is an open-label study to determine the pharmacokinetics of a new tablet formulation of GLPG1972 and to compare it with this of the liquid solution used during the First-in-Human study (GLPG1972-CL-101). The impact of food intake on the oral bioavailability of GLPG1972 administered as tablet will also be investigated in this study. A dose of 600 mg has been selected. The study is a phase I randomized open-label cross-over study with three single dose treatments:

A) 600 mg GLPG1972 oral solution after overnight fast,

B) 600 mg GLPG1972 oral tablet after overnight fast,

C) 600 mg GLPG1972 oral tablet 30 minutes after high-fat high-calorie breakfast.

A washout of at least 6 days between subsequent dosing days is respected so that no measurable plasma levels or biologically significant effects are remaining. There will be frequent assessment of adverse experiences post-dose. Twelve healthy male subjects will be selected according to the inclusion and exclusion criteria and 2 subjects each will be randomized to one of the 6 treatment sequences (ABC, ACB, BAC, BCA, CAB, CBA)

ELIGIBILITY:
Inclusion Criteria:

1. Male between 18 and 50 years of age, inclusive, on the day of signing the informed consent form (ICF).
2. A body mass index (BMI) between 18-30 kg/m², inclusive, with a weight of at least 50 kg.
3. Judged by the investigator to be in good health based upon the results of a medical history, physical examination, vital signs, 12-lead ECG, and laboratory findings.
4. Discontinuation of all medications (including over-the-counter and/or prescription medication, dietary supplements, nutraceuticals, vitamins and/or herbal supplements) except occasional paracetamol (maximum dose of 2 g/day and maximum of 10 g/2 weeks) at least 2 weeks or 5 half-lives of this medication prior to the first study drug administration. In addition, subjects must agree to follow the prohibitions and restrictions for this study.
5. Non-smokers and not be using any nicotine-containing products (abstained from smoking for at least 1 year prior to the screening).
6. Negative urine and alcohol drug screen (amphetamines, barbiturates, benzodiazepines, cannabis, cocaine, opiates, methadone, tricyclic antidepressants, and alcohol).
7. Current sexually active (and/or child wish) male agrees to use adequate contraception (see Section 4.2.4.1) from the time of first dose of study drug, during the study and until 12 weeks after the last study drug dose.
8. Subjects should be willing to consume a non-vegetarian high fat and high calorie breakfast.
9. Able and willing to sign the ICF as approved by the IEC, prior to screening evaluations

Exclusion Criteria:

1. Known hypersensitivity to study drug ingredients or a significant allergic reaction to any drug
2. Positive serology for hepatitis B virus surface antigen (HBsAg) or hepatitis C virus (HCV) or any history of hepatitis from any cause with the exception of hepatitis A.
3. History of or a current immunosuppressive condition
4. Symptoms of clinically significant illness in the 3 months before the initial study drug administration.
5. Presence or having sequelae of gastrointestinal, liver (except for Gilbert's disease) or kidney disease or other conditions known to interfere with the absorption, distribution, metabolism, or excretion of drugs.
6. History of malignancy within the past 5 years (except for basal cell carcinoma of the skin that has been treated with no evidence of recurrence).
7. Clinically relevant abnormalities detected on ECG. A first degree heart block or sinus arrhythmia will not be considered as a significant abnormality.
8. Clinically relevant abnormalities detected on vital signs.
9. Intolerance to cow milk.
10. Significant blood loss including blood donation (> 100 mL) or had a transfusion of any blood product within 12 weeks prior to the initial study drug administration.
11. Hemoglobin level below 7.5 mmol/L.
12. Treatment with any drug known to have a well-defined potential for toxicity to a major organ in the last 3 months preceding the initial study drug administration.
13. Active drug or alcohol abuse (an average intake of more than 21 glasses of wine or beer or equivalent/week) within 2 years prior to the initial study drug administration.
14. Consumption of a large quantity of coffee, tea (> 6 cups per day) or equivalent.
15. Administration of an injectable drug within 30 days prior to the initial study drug administration.

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2016-07; Primary Completion 2016-07 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Maximum observed plasma concentration (Cmax) of GLPG1972 | From pre-dose (period 1) until 6 days after the last dose (period 3)
  To study the pharmacokinetics of 600 mg GLPG1972 administered as oral liquid solution or as oral tablet after overnight fasting or administered as oral tablet after a high-fat high calorie breakfast
Plasma concentration of GLPG1972 24 hours after dosing | 24 hours after each dose
  To study the pharmacokinetics of 600 mg GLPG1972 administered as oral liquid solution or as oral tablet after overnight fasting or administered as oral tablet after a high-fat high calorie breakfast
The time of the occurrence of Cmax of GLPG1972 | From pre-dose (period 1) until 6 days after the last dose (period 3)
  To study the pharmacokinetics of 600 mg GLPG1972 administered as oral liquid solution or as oral tablet after overnight fasting or administered as oral tablet after a high-fat high calorie breakfast
The area under the plasma concentration versus time curve | From pre-dose until 6 days post-dose for each dosing period
  To study the pharmacokinetics of 600 mg GLPG1972 administered as oral liquid solution or as oral tablet after overnight fasting or administered as oral tablet after a high-fat high calorie breakfast
The apparent terminal half-life of GLPG1972 | From pre-dose (period 1) until 6 days after the last dose (period 3)
  To study the pharmacokinetics of 600 mg GLPG1972 administered as oral liquid solution or as oral tablet after overnight fasting or administered as oral tablet after a high-fat high calorie breakfast
The number of adverse events reported | From pre-dose until the Follow up (FU) visit anticipated to take place 7-10 days after the last dose
  To evaluate safety and tolerability of single oral doses of GLPG1972
Changes in clinical laboratory evaluations | From pre-dose until the Follow up (FU) visit anticipated to take place 7-10 days after the last dose
  To evaluate safety and tolerability of single oral doses of GLPG1972
Changes in vital signs | From pre-dose until the Follow up (FU) visit anticipated to take place 7-10 days after the last dose
  To evaluate safety and tolerability of single oral doses of GLPG1972
Changes in physical examination parameters | From pre-dose until the Follow up (FU) visit anticipated to take place 7-10 days after the last dose
  To evaluate safety and tolerability of single oral doses of GLPG1972
Changes in ECG parameters | From pre-dose until the Follow up (FU) visit anticipated to take place 7-10 days after the last dose
  To evaluate safety and tolerability of single oral doses of GLPG1972

CONTACTS AND LOCATIONS:
Overall Officials: Ennis Lee, MD, Study Director — Galapagos NV
Locations (1):
- PRA-EDS, Zuidlaren, Netherlands